CLINICAL TRIAL: NCT05201235
Title: Maevad - Mobilisation Active de l'Empan Visuo-Attentionel Pour la Dyslexie
Brief Title: Visual Attention Span Mobilisation for Dyslexia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Humans Matter (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-A01457-34
Record Dates: First submitted 2022-01-07; First posted 2022-01-21 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Dyslexia; Visual Attention Span Deficit
Keywords: MAEVAD; MAEVA; Reading; Remediation; Visual attention span
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Intervention Model Description: On the first group children will be trained first with MAEVAD then with a control training that does not stimulate the VA span. On contrary, on the second group children will first perform the control training and then MAEVAD.
  For each intervention the sessions will lasts 15 minutes. 5 sessions are planned per weeks for 6 weeks.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The training will be performed at home. The investigators/evaluators will send a download link of the therapy to the patient's parents without knowing which therapy it corresponds to.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MAEVAD - DeCaLigne (Experimental): The experimental group will first receive MAEVAD then the control therapy
  Interventions: Device: MAEVAD
- DeCaLigne - MAEVAD (Placebo Comparator): The control group will first receive the control therapy then MAEVAD
  Interventions: Device: DeCaLigne

INTERVENTIONS:
Device: MAEVAD — MAEVAD is a training device which aims to improve VA span as a prerequisite for learning to read. By increasing the number of distinct visual elements that can be processed simultaneously during fixation, MAEVAD is intended to improve the reading (accuracy and fluency) and spelling (lexical) performance of dyslexics who have a VA span deficit. MAEVAD is designed to be used in total autonomy by dyslexic children with a VA span disorder. The therapy takes place over 6 weeks with 5 sessions of 15 minutes per week. In order to improve compliance, the therapy has been integrated into "le Royaume d'Adelia", a serious game where the child will be able to collect materials at the end of each session that will allow him to create objects to customise a character.
  Arms: MAEVAD - DeCaLigne
Device: DeCaLigne — DéCaLigne is an intervention programme for the discovery of calculation with the number line. The objectives are to improve numerical representations in the form of a number line and to improve addition and subtraction skills. The overall principle is to move numbers or calculation results on a number line. This training does not stimulate VA span or the phonological dimensions involved in reading. This therapy is being adapted to be used in total autonomy at home and to correspond to the MAEVAD therapy in duration (5 sessions of 15 minutes per week for 6 weeks). It has also been integrated into the "royaume d'Adelia" in order to control the motivational effect of the serious game.
  Arms: DeCaLigne - MAEVAD

SUMMARY:
The aim of the study is to evaluate the efficiency of the medical device MAEVAD in improving the reading skills of children with dyslexia.

DETAILED DESCRIPTION:
MAEVAD is a digital therapy specifically designed to improve the visual attention (VA) span of children with dyslexia. Dyslexia is characterized by a specific and significant impairment in reading and/or writing production and spelling. Some profiles of children with dyslexia show a deficit in VA span, characterized by a decrease in the number of distinct visual elements that can be processed simultaneously. VA span plays a critical role in the acquisition of reading skills and specific knowledge of word spelling. Brain regions involved in visual-attentional skills are under-activated in dyslexic children with VA deficits and can be reactivated following specific and intensive VA span training.

In this study 150 children with dyslexia will be randomized in tow groups. On the first group children will be trained first with MAEVAD then with a control training that does not stimulate the VA span. On contrary, on the second group children will first perform the control training and then MAEVAD.

For each intervention the sessions will lasts 15 minutes. 5 sessions are planned per weeks for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* School children from CE2 to CM2, aged 8 to 11 years
* Dyslexic children with a VA span deficit (composite visual-attention span below the fifteenth percentile and a letter threshold above or equal to the twentieth percentile with the - - - Evadys(c) battery)
* Established diagnosis of Dyslexia
* Children whose parents/legal guardians have signed informed consent and agree to participate in the study
* Children whose first language is French or who have been educated in French since kindergarten
* Raven's Progressive Matrices score above the 20th percentile or a WISC IV or V Verbal Comprehension Index or WISC IV or V Perceptual/Fluid Reasoning Index above 85 or documented/objectifiable absence of intellectual deficit
* Child with access to a computer
* Normal or corrected vision and audition

Exclusion Criteria:

* Attention deficit hyperactivity disorder,dysphasia, dyspraxia, Autism Spectrum Disorder
* Neurological disorders
* Children who have missed 3 months or more of school in the current or previous year (excluding lockdown)
* Children not affiliated to a social security scheme

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-07-05 (Actual)

PRIMARY OUTCOMES:
Reading speed | 10 weeks to baseline
  Measure of reding time from texts of 122 to 152 words
Reading speed | 18 weeks to baseline
  Measure of reding time from texts of 122 to 152 words
Reading speed | 26 weeks to baseline
  Measure of reding time from texts of 122 to 152 words

SECONDARY OUTCOMES:
Reading skills | 10 weeks to baseline
  Word and pseudoword reading tests (reding time and accuracy) Text reading (reading time and accuracy)
Reading skills | 18 weeks to baseline
  Word and pseudoword reading tests (reding time and accuracy) Text reading (reading time and accuracy)
Reading skills | 26 weeks to baseline
  Word and pseudoword reading tests (reding time and accuracy) Text reading (reading time and accuracy)
Orthographic skills | 10 weeks to baseline
  Lexical-spelling judgment (Accuracy and time) Words and pseudowords dictation (Accuracy)
Orthographic skills | 18 weeks to baseline
  Lexical-spelling judgment (Accuracy and time) Words and pseudowords dictation (Accuracy)
Orthographic skills | 26 weeks to baseline
  Lexical-spelling judgment (Accuracy and time) Words and pseudowords dictation (Accuracy)
VA Span | 10 weeks to baseline
  Evadys test : EVADYS(c) provides a reliable diagnosis of visual-attention span disorder. The software includes three versions of the global and partial report tests, each adapted to a given age group.
VA Span | 18 weeks to baseline
  Evadys test : EVADYS(c) provides a reliable diagnosis of visual-attention span disorder. The software includes three versions of the global and partial report tests, each adapted to a given age group.
VA Span | 26 weeks to baseline
  Evadys test : EVADYS(c) provides a reliable diagnosis of visual-attention span disorder. The software includes three versions of the global and partial report tests, each adapted to a given age group.
Phonologic skills | 10 weeks to baseline
  Evalec(c) test : The child will have to delete, orally, the first phoneme of the pseudowords presented on the screen.
  12 pseudowords with a consonant-vowel-consonant structure and 12 with a consonant-consonant-vowel structure are presented one by one on the screen.
Phonologic skills | 18 weeks to baseline
  Evalec(c) test : The child will have to delete, orally, the first phoneme of the pseudowords presented on the screen.
  12 pseudowords with a consonant-vowel-consonant structure and 12 with a consonant-consonant-vowel structure are presented one by one on the screen.
Phonologic skills | 26 weeks to baseline
  Evalec(c) test : The child will have to delete, orally, the first phoneme of the pseudowords presented on the screen.
  12 pseudowords with a consonant-vowel-consonant structure and 12 with a consonant-consonant-vowel structure are presented one by one on the screen.
Mathematical skills | 10 weeks to baseline
  DeCaLigne(c) and Examath(c): The child will have to find the position of a number on a numerical line and answer mental calculation.
Mathematical skills | 18 weeks to baseline
  DeCaLigne(c) and Examath(c): The child will have to find the position of a number on a numerical line and answer mental calculation.

CONTACTS AND LOCATIONS:
Overall Officials: Mélodie FOUILLEN, PhD, Study Chair — Humans Matter
Locations (55):
- France (55):
  - MARTINELLI Karen, Ajaccio
  - BERARD Marine, Albertville
  - CARCEY-CADET Elise, Albertville
  - KOUASSI-PUJOL Marie, Albi
  - CLAVIER-MARCOUX Laetitia, Antibes
  - BOCCOGNANI Jordane, Argences en Aubrac
  - CHAUVET Clémence, Arles
  - CHABERT Claire, Bagnères-de-Bigorre
  - SCHMITT Véronique, Biganos
  - CRABÉ Marion, Billère
  - BIRAN Sandrine, Bordes
  - VALLERY Théoline, Brest
  - LADOUL Marine, Brive-la-Gaillarde
  - COURANT Sabrina, Cabasse
  - CONTESTI Véronique, Champagne-au-Mont-d'Or
  - MINIAC-FOURNIER Stéphanie, Château-Gontier
  - CASTERES Catherine, Digoin
  - PASQUIER Amélie, Fay-de-Bretagne
  - LEGENDRE Laure, Fontenay-sous-Bois
  - FORTIER Anne, Garches
  - BLANC Emilie, Givors
  - KRAYEM Mona, Guichainville
  - RIZK Joumana, Guichainville
  - SHAW PERRIN Anne-Sophie, Irigny
  - DE MUYNCK Solène, Lamballe
  - CADALEN Hélène, Lanmeur
  - VOLUET FROMENT Adeline, Le Chesnay
  - BERNARD-DENIS Fabienne, Le Havre
  - TERRASSON Cécile, Le Touquet-Paris-Plage
  - CALAIS Cécile, Liancourt
  - Britt, Lux
  - GOBÉ Valérie, Machecoul
  - JORDANIS Mélanie, Marignier
  - VERLOT-MORY Ludivine, Meuilley
  - MAZERAN Anne-Cécile, Miribel
  - KIS Nathalie, Montigny-le-Bretonneux
  - EMERIAU Mathilde, Nantes
  - LHUILLIER Françoise, Neufchâteau
  - LEJOSNE Julie, Paimpol
  - BRESSON Raphaëlle, Plaisir
  - BERTHELOT Florence, Plérin
  - BERTHOLOM Anne-Marine, Ploudalmézeau
  - ZIMMERMAN Amélie, Remoulins
  - CAMUS-BRUNEAU Anne, Rezé
  - KOCHEL Jeanne-Marie, Saint-Germain-en-Laye
  - VIERLING Pauline, Saint-Leu
  - LECLERC LE COADOU Rozenn, Saint-Lô
  - NADAUD Stéphanie, Saint-Nom-la-Bretêche
  - REVERSE Christelle, Saint-Péray
  - DESCENDRE Myriam, Saint-Quentin
  - RAYNAUD LEGROS Caroline, Sainte-Anne
  - AÏT LEMKADEM Mimouna, Sartrouville
  - FRITSCH Colombine, Schiltigheim
  - CARRIQUE Pascale, Tourrettes
  - KALCK Christine, Vendenheim

IPD SHARING:
Plan to Share IPD: No